CLINICAL TRIAL: NCT06290401
Title: A Socio-ecological Approach for Improving Self-management in Adolescents With SCD
Acronym: SC-Thrive
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Nemours Children's Health System (Other); Emory University (Other); Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023-0671
Record Dates: First submitted 2024-02-15; First posted 2024-03-04 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Anemia, Sickle Cell
Keywords: adolescent and young adult (AYA); self-management; behavioral intervention; sickle cell disease
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Intervention Model Description: Participants will be allocated to SCThrive or SCHealthED (uniform standard care) using a randomized block design for age group (13-17 years of age or 18-21 years of age) with a predefined block size of 4.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Investigator and Outcomes assessors will not know the condition to which participants have been randomized.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Treatment (Active Comparator): SCThrive is a virtual, 8-week, virtual group-based, behavioral self-management intervention that includes daily use of a companion mobile app.
  Interventions: Behavioral: SCThrive
- Control Condition (Placebo Comparator): Participants randomized to SCHealthED will receive usual care plus 7 text messages consisting of SCD educational facts to ensure the care is uniform across sites.
  Interventions: Other: SCHealthED

INTERVENTIONS:
Behavioral: SCThrive — SCThrive is a virtual, 8-week, virtual group-based, behavioral self-management intervention that includes daily use of a companion mobile app.
  Arms: Active Treatment
Other: SCHealthED — Standard of care plus 7 SCD educational text messages to ensure education is uniform across sites
  Other Names: Uniform Standard Care
  Arms: Control Condition

SUMMARY:
The goal of this clinical trial is to evaluate the impact of SCThrive (a behavioral self-management intervention) on patient activation, self-management behaviors, daily functioning, and emergency room visits in 260 adolescents and young adults with sickle cell disease (SCD) ages 13-21 receiving care at 1 of 4 pediatric SCD clinics.

The main question[s]it aims to answer are:

* Does SCThrive improve patient activation?
* Does SCThrive improve self-management behaviors, daily functioning, and decrease emergency room visits?
* Are any improvements maintained 3 months after treatment?

Participants will complete self-management related surveys before, after, and 3 months following their participation in an 8- week, virtual group intervention with an accompanying mobile app (SCThrive).

Researchers will compare outcomes for participants who receive SCThrive and participants who receive uniform standard care (SCHealthED which = standard of care plus SCD educational text messages) to see if there are differences in patient activation, self-management behaviors, daily functioning, and emergency room visits.

DETAILED DESCRIPTION:
The research team's pilot work demonstrated improved patient activation (knowledge, skills, and self-efficacy) and self-management behaviors in adolescents and young adults (AYA) with sickle cell disease (SCD) compared to a control condition. Further analyses revealed that participants who used the app more frequently showed greater improvements. Thus, this study will maximize the clinical benefit of SCThrive by 1) adding app engagement strategies, 2) conducting a more systematic assessment of barriers including social contributors to health, and 3) integrating ways to address these barriers into the intervention.

Study Aims: The aims are to examine the impact of SCThrive on patient activation (primary outcome; Aim 1) and self-management behaviors, daily functioning, and emergency room visits (secondary outcomes) at post-treatment and follow-up (Aim 2). It is hypothesized that adolescents randomized to SCThrive will have greater improvement in patient activation (primary outcome) compared to those randomized to uniform standard care (control condition). The research team will also explore the relationship between social determinants of health (SDOH)-related barriers (e.g., stigma, access to care) and treatment response (i.e., patient activation and self-management behaviors).

ELIGIBILITY:
Inclusion Criteria:

* Patient of a participating SCD Clinic
* Confirmed diagnosis of SCD
* 13-21 years of age

Exclusion Criteria:

* Another chronic disease (which would complicate measurement of patient activation)
* Non-English-speaking
* Cognitive or psychiatric disorder that the physician or study therapists believe would impair study participation.

Ages: 13 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 310 (Estimated)
Dates: Start 2025-02-03 (Actual); Primary Completion 2028-01-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Patient Activation | baseline, up to 4 weeks after treatment ends, 3 to 4 months after treatment ends
  Self-reported patient activation as measured by the Patient Activation Measure -13 (PAM-13), which is a 13 item measure on skills, knowledge, confidence and readiness for self-management developed by Hibbard et al., 2005. Items are rated on a 4-point Likert scale of 1 = "Disagree Strongly" to 3 = "Strongly Agree." Raw scores range from 13 to 52 and are converted to scores that range from 0 to 100. This score was then divided into four levels of activation, which reflect a developmental progression from being passive with regard to one's health to being proactive: Level 1 (score of 0.0 - 47.0), Level 2 (47.1 - 55.1), Level 3 (55.2 - 72.4), and Level 4 (72.5 - 100). Higher scores indicate more behavioral activation.

SECONDARY OUTCOMES:
Self-Management Behaviors | baseline, up to 4 weeks after treatment ends, 3 to 4 months after treatment ends
  self-reported self-management behaviors as measured by the Transition Readiness Assessment Questionnaire - 6 (TRAQ-6), which is a well-validated 20-item questionnaire that measures the skills needed to manage a chronic condition independently. Items are rated on a 5-point Likert scale of 1 = "No, I do not know how" to 5 = "Yes, I always do this when I need to" and divided into 5 subscales: Managing Medication, Appointment Keeping, Tracking Health Issues, Talking with Providers, and Managing Daily Activities. Overall and subscale scores are calculated by averaging the scores of answered items. Mean scores range from 1 to 5 with higher scores indicating better self-management.
Daily Functioning | baseline, up to 4 weeks after treatment ends, 3 to 4 months after treatment ends
  The Functional Disability Inventory is a self-report measure of limitations in children's physical and psychosocial functioning due to their physical health. The instrument consists of 15 items concerning activity limitations due to "being sick or not feeling well" during the past 2 weeks. Total scores ranging from 0 to 60 are computed by summing the ratings for each of the 15 items on the FDI. Higher scores indicate greater perceived functional disability.
Emergency Room (ER) Visits | 6 months prior to treatment; 6 months post-treatment
  number of emergency room visits
Self-Management Skills | baseline, up to 4 weeks after treatment ends, 3 to 4 months after treatment ends
  Participants complete the UNC TRxANSITION Scale, an interview administered by trained independent evaluators to measure the skills of youth with chronic conditions. For this study, we will administer 6 of the 10 possible subscales: Type of Chronic Health Condition, Medications, Adherence, Nutrition, Self-Management Skills, and New Health Care Providers. Each item is scored individually as either 1 (adequate knowledge/skill mastery), 0.5 (some knowledge/skill attainment), or 0 (no knowledge/skill attainment). Higher scores indicate better self-management. Subscale scores are calculated by dividing the patient's score by the total possible subscale score. Subscale scores are then combined to create a total score, ranging from 0 to 10, but since we will only use 6 scales, 0 to 6. Total and subscale proportion scores will be used in analyses.
Health-related quality of life | baseline, up to 4 weeks after treatment ends, 3 to 4 months after treatment ends
  Patient report of sickle cell disease (SCD)-specific quality of life (QOL) and pain, as measured by the Pediatric Quality of Life (PedsQL) SCD Module, which assesses several domains of health-related quality of life (HRQOL), including pain impact, fatigue, pain management, emotions, communication, and treatment adherence. Total score only. Scores range from 0 to 100, with higher scores indicating higher HRQOL or higher functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Lori E. Crosby, PsyD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (4):
- United States (4):
  - Nemours Children's Health, Wilmington, Delaware
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No
Only de-identified data will be shared with other researchers. Deidentified data sets will be available on the Open Science Framework.